CLINICAL TRIAL: NCT06507306
Title: A Phase 1/1b, Open-label, Multicenter, Dose Escalation and Dose Expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of KQB198 as Monotherapy and in Combination With Anti-cancer Agents in Participants With Advanced Solid Malignancies
Brief Title: A Study to Investigate the Safety and Efficacy of KQB198 as Monotherapy and in Combination in Participants With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kumquat Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQB198-101
Record Dates: First submitted 2024-07-01; First posted 2024-07-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — osimertinib; amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Monotherapy Dose Escalation (Experimental)
  Interventions: Drug: KQB198
- Combo Therapy Dose Escalation (Experimental)
  Interventions: Drug: KQB198; Drug: Osimertinib; Drug: Amivantamab
- Combo Therapy Dose Expansion - RP2D (Experimental)
  Interventions: Drug: KQB198; Drug: Osimertinib; Drug: Amivantamab
- Combo Therapy Dose Expansion - RP2D-1 (Experimental)
  Interventions: Drug: KQB198; Drug: Osimertinib; Drug: Amivantamab
- Combo Therapy Dose Expansion OBD (Experimental)
  Interventions: Drug: KQB198; Drug: Osimertinib; Drug: Amivantamab

INTERVENTIONS:
Drug: KQB198 — Oral KQB198
Drug: Osimertinib — Oral Osimertinib
  Other Names: Tagrisso
  Arms: Combo Therapy Dose Escalation; Combo Therapy Dose Expansion - RP2D; Combo Therapy Dose Expansion - RP2D-1; Combo Therapy Dose Expansion OBD
Drug: Amivantamab — Subcutaneous administration
  Arms: Combo Therapy Dose Escalation; Combo Therapy Dose Expansion - RP2D; Combo Therapy Dose Expansion - RP2D-1; Combo Therapy Dose Expansion OBD

SUMMARY:
The goal of this clinical trial is to learn if KQB198 works to treat advanced solid tumor cancer in adults. It will also learn about the safety of KQB198. The main questions it aims to answer are:

* What is the safe dose of KQB198 by itself or in combination with other anti-cancer drugs?
* Does KQB198 alone or in combination with other anti-cancer drugs decrease the size of the tumor?
* What happens to KQB198 in the body?

Participants will:

* Take KQB198 daily, alone or in combination with another anti-cancer drug
* Visit the clinic about 8 times in the first 8 weeks, and then once every 4 weeks after that

ELIGIBILITY:
Inclusion Criteria:

* PART 1 - Histologically confirmed diagnosis of a solid tumor malignancy with any of the following oncogenic mutations: EGFR, RAS, PTPN11, or SOS1 mutations, or inactivating mutations of NF1.
* PART 1 - (Osimertinib and Amivantamab arms) and Part 2 Cohort A and Cohort B: Histologically confirmed diagnosis of NSCLC with activating EGFR mutation and progression on osimertinib
* Part 3 - Cohort A: Histologically confirmed diagnosis of NSCLC with exon 20 insertion EGFR mutation
* Unresectable or metastatic disease
* No available treatment with curative intent
* Adequate organ function
* Measurable disease per RECIST 1.1.

Exclusion Criteria:

* Prior therapy with a similar mechanism of action to KQB198
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions likely to alter absorption of study treatment or result in inability to swallow
* History of interstitial lung disease
* Cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experience treatment-emergent adverse events, serious adverse events, and dose-limiting toxicities (Part 1) | 28 Days
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of AEs, SAEs, and DLTs, from first dose of study treatment to 28 days after last dose of study treatment.
Recommended Phase 2 Dose (RP2D) (Part 1) | up to 30 months
  Evaluate safety and assess number of patients with dose-limiting toxicity to determine the RP2D.
Efficacy and Optimal Biologic Dose of study treatment, as measured by Objective Response Rate (ORR) (Parts 2 and 3) | up to 30 months
  Objective response is the proportion of subjects that experience confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 during the time period from 1st dose of study treatment until last dose.

SECONDARY OUTCOMES:
Concentration-time curve (AUC) | up to 30 months
Maximum plasma concentration (Cmax) | up to 30 months
Time to maximum plasma concentration (tmax) | up to 30 months
Overall survival (OS) | up to 30 months
Progression-free survival (PFS) | up to 30 months
Overall response rate (ORR) | up to 30 months
Duration of response (DOR) | up to 30 months
Time to response (TTR) | up to 30 months

CONTACTS AND LOCATIONS:
Locations (35):
- United States (10):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Sarah Cannon Research Institute at Florida Cancer Specialists - Lake Nona -, Orlando, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Henry Ford Health System, Detroit, Michigan
  - David H. Koch Center for Cancer Center at Memorial Sloan Kettering Cancer Center, Long Island City, New York
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - New Experimental Therapeutics of San Antonio - NEXT Oncology, San Antonio, Texas
  - New Experimental Therapeutics of Virginia - NEXT Oncology, Fairfax, Virginia
- France (5):
  - Institut Paoli-Calmettes, Marseille, Bouches-du-Rhône
  - Institut de Cancerologie de l'Ouest - site St-Herblain, Saint-Herblain, Loire-Atlantique
  - CHU Bordeaux - Hopital Saint-Andre, Bordeaux, Nouvelle-Aquitane
  - IUCT-Oncopole, Toulouse, Occitaine
  - CHU de Nantes - Hopital Nord Laennec, Nantes, Pays de la Loire Region
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome, Lazio
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
- Spain (10):
  - Hospital Universitari Quiron Dexeus Barcelona, Barcelona, Catalonia
  - Hospital Universitario Vall d'Hebron, Barcelona, Catalonia
  - New Experimental Therapeutics (NEXT) Oncology Barcelona, Barcelona
  - South Texas Accelerated Research Therapeutics (START) Barcelona- HM Nou Delfos, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - South Texas Accelerated Research Therapeutics (START) Madrid - CIOCC, Madrid
  - New Experimental Therapeutics (NEXT) Oncology Madrid - Hospital Quironsalud Madrid, Madrid
  - South Texas Accelerated Research Therapeutics (START) Madrid - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Quirónsalud Málaga, Málaga
  - Clinica Universidad de Navarra - Pamplona, Pamplona
- Taiwan (4):
  - Chi-Mei Hospital - Liouying Branch, Liuying, Tainan City
  - National Taiwan University Hospital, Taipei, Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei